CLINICAL TRIAL: NCT03713151
Title: Feasibility of a Blended Therapy Approach: Face-to-face Physiotherapy Sessions Combined With an Interactive Tablet-based Exercise Program for People With Rare Diseases.
Brief Title: Feasibility of a Blended Therapy Approach
Acronym: bletheRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00970
Record Dates: First submitted 2018-08-29; First posted 2018-10-19 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Telemedicine; Exercise; Feasibility; Myositis; Haemophilia
Keywords: Telemedicine, Feasibility, Exercise
MeSH Terms: conditions — Motor Activity; Myositis; Hemophilia A

STUDY DESIGN:
Intervention Model Description: Feasibility study with a pre-post comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dividat FIT: Computer based exercise (Experimental): One arm with 10-15 Haemophilia patients and 10-15 Myositis patients.
  Interventions: Other: Dividat FIT

INTERVENTIONS:
Other: Dividat FIT — The study intervention is a blended therapy approach of face-to-face physiotherapy sessions with an interactive tablet-based home exercise program.

SUMMARY:
Exercise is an important part of therapy guidelines in the rehabilitation of rare diseases (RDs) as Haemophilia and Myositis. The aim of this study is not to evaluate a new therapy intervention, but to evaluate the delivery of this intervention. In clinical practice, patients are usually instructed to perform an exercise program at home. Normally, a physiotherapist (PT) provides an instruction (paper-) sheet. In this study, the investigators evaluate the feasibility of an interactive tablet-based way of delivery. The exercise program is - as usual in physiotherapy - individually tailored by the PT.

DETAILED DESCRIPTION:
Myositis and haemophilia belong with a prevalence rate of 0.4-17.3 of 100'000 and 2-12 of 100'000, respectively to the group of RDs. The fact that a RD affects only a small number of people, indicates that rehabilitation knowledge outside the specialised medical centers is rare. Thus, since many people with RD do not live nearby these institutions, they do not have direct acces to rehabilitation programmes. The University Hospital Zurich (USZ) offers medical treatment and Rehabilitation Support in such reference centers, among others for people with myositis (PWM) and for people with haemophilia (PWH).

Although these two diseases differ strongly in their underlying cause, affected persons are confronted with similar problems: PWM and PWH suffer from musculoskeletal problems and therefore, a physically active lifestyle is essential to maintain good health. Nevertheless, PWM and PWH were previously discouraged from participating in physical exercise. Consequently, both groups are less physically active, have a lower fitness level and a higher risk for comorbidities, compared to healthy people. Nowadays, the beneficial effects of exercise in PWH and in PWM are well accepted and there is evidence that PWH and PWM profit from physical exercise programs.

Despite the encouraging benefits of physical exercise in PWH and PWM, these may be challenged with more barriers to start and maintain an exercise program, compared to healthy persons, e.g. due to reduced accessibility of specialised physiotherapists.

Telerehabilitation (TR), a subfield of telemedicine, may help to overcome some of the barriers to exercise regularly and connect PWH/PWM with specialised physiotherapists. TR is defined as the provision of rehabilitation services from a distance using telecommunication technologies as the delivery medium. This approach may optimize the timing, intensity and sequencing of interventions and provide opportunities for individuals to receive rehabilitation in their own social and professional environments from disease-specialised caregivers. An additional advantage of TR is the possibility to implement different persuasive technologies such as personalisation, self-monitoring, tailoring, goal setting, comparison and conditioning through positive and negative reinforcement in the development of exercise programmes. These technologies help to make exercise programmes more enjoyable and, therefore, enhance patients' motivation to exercise regularly.

Furthermore, the importance of individual and social support has been emphasized in several reviews evaluating health behaviour change for example becoming more active. This kind of support can be integrated in the design of a TR program and it can further be enhanced by blending TR with face-to-face sessions. The so-called blended therapy is a promising approach combining the advantages from traditional rehabilitation and new technologies.

The aim of this study is to evaluate feasibility of a blended therapy approach, combining a tablet-based exercise program, called "Dividat Fit" with face-to-face therapy sessions for PWH and PWM.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of mild Haemophilia or Myositis

* able to walk 20 meters without walking aids
* currently exercising less than one training session per week (training = vigorous activity)
* maintenance of a stable medical regimen for 4 weeks prior to initiation of study and considered to maintain a stable regimen for the course of the study
* signed informed consent to participate in the study

Exclusion Criteria:

* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, severe cardiovascular and/or pulmonary disease, severe osteoporosis, pulmonary hypertension, pain syndrome, paresis)
* Contraindications to physical exercise for People with Haemophila: Factor-prophylaxis-regimen, inhibitor positive, less than 6 months after arthroplasty surgery, acute joint or muscle bleeding within the last 30 days for People With Myosites: acute exacerbation of inflammation
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Known pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited in the study | Will be assessed approximately 6 months after start of study
  Recruitment rate, reasons for denial and exlusion and drop-outs

SECONDARY OUTCOMES:
Adherence to the "Dividat Fit" exercise program | Will be assessed approximately 6 months after start of study
  Number of completed training sessions
Perceived usefulness and perceived ease of use of Dividat Fit | 10 Minutes for each patient after the end of the 12-week intervention program
  Technology Assessment Model Questionnaire : 7-point Likert scale ranging from "strongly disagree" (rated as 1) to "strongly agree" (rated as 7). The TAM model can explain the users' motivation by three factors in subscales: perceived ease of use, perceived usefulness and attitude toward using the Technology.
Perceived satisfaction of Dividat FIT | 10 Minutes for each patient after the end of the 12-week intervention program
  Satisfaction Questionnaire : 5-point Likert scale ranging from "strongly agree" (rated as 1) to "strongly disagree" (rated as 5). The model can explain the users' satisfaction rating by following factors in subscales: Satisfaction of physiotherapy sessions, satisfaction of the home program, satisfaction of the technical aspects and aspects that improved the motivation for the computer exercise program.
Hand-held dynamometry | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  Isometric Muscle Force
Manual Muscle testing | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  MMT8 only for People with Myosites
Expanded Timed Get-up-and-Go | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  ETGUG
30 second chair stand | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  Chair raise
30 second arm curl | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  lift a 1 kg weight above the head until the elbow is fully extended in a 30 second period at a comfortable pace
Functional Index 2 Test (FI2) : Number of repetitions for muscle endurance | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  In the FI2 test, patients perform as many repetitions for the subscales schoulder flexion, shoulder abduction, head lift, hip flexion, step test, heel lift and toe lift at a standardised movement pace untill a maximal number of correct repetitions is reached (60 repetitions for shoulder flexion, shoulder abduction, head lift, hip flexion and step test and 120 repetitions for heel lift and toe lift).If the patient cannot keep up the pace or perform the correct movement, then the amount of the correctly performed repetitions for a subscale is noted.
Stanford Health Assessment Questionnaire Disability Index (HAQ) | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  The HAQ consists of 20 questions divided into eight subscales on a 4 Point likert scale: Dressing, rising, eating, walking, hygiene, reaching, grip function, and performing activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). The summed subscores are divided by 8, to receive the total score.
Health related disability and quality of life (SF-36) | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  The SF-36 is a generic patient-reported outcome measure aimed at quantifying health related quality of life (HRQOL). The SF-36 includes 36 questions divided in eight subscales: Limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being), limitations in usual role activities because of emotional problems, vitality (energy and fatigue), general health perceptions. The eight subscales can be divided into two main components: physical component summary (PCS) and mental component summary (MCS). In the two main components higher scores indicate better HRQOL.
Myositis Activity Profile questionnaire (MAP) | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  The MAP includes 32 items which can be answered on a 7-point Likert scale; where 1= no difficulty to perform and 7= impossible to perform. These items are divided into four subscales (movement activities, activities of moving around, personal care, and domestic activities) and four single items (keeping in touch with close friends and relatives, avoiding overexertion during daily activities, being able to cope with work and/or housework to a satisfactory degree, and being able to do recreational activities of choice).
Haemophilia & Exercise Project-Test-Questionnaire (HEP-Test-Q) | Measurement approximately, two weeks before the start of the exercise intervention and after the end of the 12-week intervention program.
  The HEP-Test-Q is a questionnaire, assessing subjective physical performance of patients with haemophilia. It consists of 25 items pertaining to four domains "mobility", "strength & coordination", "endurance" and "body perception" and one single item, which assesses changes in physical functioning in comparison to the previous year. Each item can be answered on a 5-point ordinal scale varying from 1 (never) to five (always).

CONTACTS AND LOCATIONS:
Overall Officials: Ruud Knols, PhD, Principal Investigator — University of Zurich
Locations (1):
- Ruud Knols, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pfister PB, Knols RH, de Bie RA, de Bruin ED. Feasibility of a blended therapy approach in the treatment of patients with inflammatory myopathies. Arch Physiother. 2021 May 27;11(1):14. doi: 10.1186/s40945-021-00108-z. PMID 34039438